CLINICAL TRIAL: NCT06756269
Title: A Randomised, Double-blind, Placebo and Positive Controlled, Phase 2 Clinical Trial to Evaluate the Safety and Immunogenicity of 15-valent Human Papillomavirus Recombinant Vaccine (Hansenulapolymorpha) in Healthy Chinese People Aged 9-45 Years
Brief Title: To Evaluate the Safety and Immunogenicity of 15-valent HPV Recombinant Vaccine in Chinese People Aged 9-45 Years
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 15-HPV-2001
Record Dates: First submitted 2024-12-31; First posted 2025-01-01 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: HPV Infection; HPV-Related Carcinoma; HPV-Related Intraepithelial Neoplasia; Genital Wart
MeSH Terms: conditions — Papillomavirus Infections; Condylomata Acuminata

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Medium dose for 15-HPV vaccine (Experimental): Participants aged 9-45 years were given 3 doses of medium dose 15-HPV vaccine intramuscular into the upper arm deltoid muscle according to 0, 2, and 6 months immunization schedule
  Interventions: Biological: Medium dose for 15-HPV vaccine
- High dose for 15-HPV vaccine (Experimental): Participants aged 9-45 years were given 3 doses of high dose 15-HPV vaccine intramuscular into the upper arm deltoid muscle according to 0, 2, and 6 months immunization schedule
  Interventions: Biological: High dose for 15-HPV vaccine
- Placebo (Placebo Comparator): Participants aged 9-45 years were given 3 doses of placebo intramuscular into the upper arm deltoid muscle according to 0, 2, and 6 months immunization schedule
  Interventions: Biological: Placebo
- 9-HPV-vaccine (Active Comparator): Participants aged 18-45 years were given 3 doses of 9-HPV vaccine intramuscular into the upper arm deltoid muscle according to 0, 2, and 6 months immunization schedule
  Interventions: Biological: 9-HPV vaccine

INTERVENTIONS:
Biological: Medium dose for 15-HPV vaccine — Participants aged 9-45 years were given 3 doses of medium dose 15-HPV vaccine intramuscular into the upper arm deltoid muscle according to 0, 2, and 6 months immunization schedule
  Arms: Medium dose for 15-HPV vaccine
Biological: High dose for 15-HPV vaccine — Participants aged 9-45 years were given 3 doses of high dose 15-HPV vaccine intramuscular into the upper arm deltoid muscle according to 0, 2, and 6 months immunization schedule
  Arms: High dose for 15-HPV vaccine
Biological: Placebo — Participants aged 9-45 years were given 3 doses of placebo intramuscular into the upper arm deltoid muscle according to 0, 2, and 6 months immunization schedule
  Arms: Placebo
Biological: 9-HPV vaccine — Participants aged 9-45 years were given 3 doses of 9-HPV vaccine intramuscular into the upper arm deltoid muscle according to 0, 2, and 6 months immunization schedule
  Arms: 9-HPV-vaccine

SUMMARY:
To evaluate the safety and Immunogenicity of 15-valent HPV vaccine in 9-45year-old participants.

DETAILED DESCRIPTION:
A Randomized, double-blind, placebo and positive controlled trial is planned in 330 healthy participants across two age groups (18-45 years and 9-17 years) to evaluate the safety and immunogenicity of the 15-valent HPV vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 9-45；
2. Participants aged 18-45 who can provide legal identification，participants aged 9-17 and their guardian can provide legal identification；
3. Participants and/or their guardian sign an informed consent form;
4. Axillary temperature less than 37.3 ℃（>14 years old）or less than 37.5℃（≤14 years old）at the time of enrollment；
5. Be able to comply with study protocol requirements；
6. Women with reproductive age take effective contraceptive measures within 2 weeks before enrollment in the study, and were not pregnant at the time of enrollment (negative blood pregnancy test), did not have lactation period, and had no birth plan within the 30 days after receiving the whole vaccination;
7. Agree to take effective contraceptive measures within 30 days after receiving the whole vaccination (effective contraceptives include: oral contraceptives, injection or embedding contraceptives, sustained release topical contraceptives, hormone patches, intrauterine devices), sterilization, abstinence, condoms (male), diaphragms, cervical caps, etc.

Exclusion Criteria:

1. Have been vaccinated with other HPV vaccines or planned to vaccinate other HPV vaccines during the study period；
2. Plan to participate other clinical trials during the study period，or participated other clinical trials （including vaccine or drug）and received medication or vaccine within 3 months before enrollment ,
3. History of positive HPV testing (including types not covered by the trial vaccine) among the participants aged 18-45 years old;
4. History of CIN2/AIS/Cervical Cancer/Pelvic radiation therapy in female participants;
5. History of HPV-related external genital diseases (such as genital warts, Vulvar intraepithelial neoplasia, Vaginal intraepithelial neoplasia, Penis/perianal/perineum intraepithelial neoplasia, Penile/perianal/perineal cancer) 、anal intraepithelial neoplasia and related cancer, or head and neck cancer；history of sexually transmitted diseases (including syphilis， Gonorrhea, genital chlamydia infection, genital herpes, soft chancre, sexually transmitted lymphogranuloma, inguinal granuloma, etc.);
6. Has been diagnosed as having congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection/AIDS, SCID; Or Autoimmune Diseases (such as systemic lupus erythematosu, Rheumatoid arthritis, juvenile Rheumatoid arthritis, Pernicious Anemia, Ulcerative colitis, Type 1 diabetes, Graves' disease, hashimoto thyroiditi, etc.);
7. History of convulsions, epilepsy, except of febrile convulsions in children 5 years of age and younger;
8. History of severe allergy that requires medical intervention, including but not limited to severe adverse reactions caused by vaccine or drug, eg anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenia sexual purpura, local allergic necrosis (Arthus reaction), widespread urticaria, dyspnea, angioedema, etc.; History of severe side effect caused by vaccination or severe allergy to any of the components of the investigational vaccine, including histidine, sodium chloride, aluminium phosphate, Polysorbate 80 and water for injection;
9. Severe diseases, as determined by the investigator, that affect vaccination eligibility, whether past or current, include severe cardiovascular disease, severe liver and kidney disease, malignant tumor, and serious infectious disease, such as: tuberculosis, viral hepatitis, etc.;
10. Before the enrollment, the physical examination was untreatment or uncontrolled hypertension, (18-45 year old: systolic blood pressure ≥140mmHg and / or diastolic blood pressure ≥90mmHg, 9-17 year old: systolic blood pressure ≥120mmHg and / or diastolic blood pressure ≥80mmHg);
11. Coagulation disorders: such as Congenital or acquired hemophilia, Coagulation factor deficiency, clotting disorders, thrombocytopenia, etc.;
12. No spleen or functional spleen, and no spleen caused by any condition;
13. Receive any Immunosuppressive therapy product within 1 month prior to the first vaccination, or plan to receive such product from Day 0 to Month 7 (30 days after receiving the third dose of vaccination)，e.g. systemic medication for glucocorticoid (>20mg/day or 2mg/kg/day, continuous use ≥2 weeks), but local medication can be used (such as ointment, eye drops, inhalants) Or nasal spray);
14. Receive any immunoglobulin or blood product within 3 months prior to the first injection, or plan to receive such product from Day 0 to Month 7 (30 days after receiving the third dose of vaccination);
15. 3 days before vaccination, suffering from acute illness or acute exacerbation of chronic disease; using fever reducer, Antihistamines, and Analgesics(such as: Acetaminophen, Ibuprofen, loratadine, Cetirizine, etc. )
16. Receiving inactivated vaccine or recombinant vaccine or live-attenuated vaccine or nucleic acid vaccine or adenovirus vaccine within 14 days before vaccination;
17. History of mental disorders or family history of mental health disorder (immediate family);
18. Plan to move out of the city before the end of the study or leave the local area for a long time during the scheduled study visit;
19. The investigator believes that the participant has any condition that may interfere with the assessment of the purpose of the study.

Ages: 9 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 330 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2026-01-13 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Up to 30 minutes after any vaccination
  AE of local and systemic reactions within 30 minutes after each dose
Percentage of Participants With Solicited Adverse Events | Up to 14 days after any vaccination
  The percentage of participants with one or more solicited AEs was assessed.
Percentage of Participants With Unsolicited Adverse Events | Up to 30 days after any vaccination
  Percentage of Participants With Unsolicited Adverse Events
Percentage of Participants With Serious Adverse Events | From Day 0 after the first dose of vaccination to 6 months after the thrid dose
  The percentage of participants with one or more SAEs was assessed
Percentage of Female Participants With Pregnancy Events | From Day 0 after the first dose of vaccination to 6 months after the thrid dose
  The percentage of participants with Pregnancy Events was assessed

SECONDARY OUTCOMES:
Immunogenicity after receiving 3 doses of 15-HPV vaccine | Up to 31 days after the third vaccination
  Geometric mean titer (GMT) of anti-vaccine containing corresponding type of neutralizing antibody in subjects aged 18-45 years on the 31-day after the third dose of immunization
Immunogenicity of 15-HPV vaccine | Up to 31 days after the third vaccination
  Seroconversion rate （SCR）of the anti-vaccine containing the corresponding type of neutralizing antibody on day 31 after total immunization in subjects aged 18-45 years
Immunogenicity after receiving 3 doses of 15-HPV vaccine among the participants | Up to 31 days after the third vaccination
  Geometric Mean Fold Increase (GMI) and 4-fold increase rates of anti-vaccine corresponding types of neutralizing antibodies in baseline seropositive subjects aged 18-45 years at day 31 after immunization

CONTACTS AND LOCATIONS:
Overall Officials: Yi Mo, Master, Principal Investigator — Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention
Locations (1):
- Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No